CLINICAL TRIAL: NCT03229447
Title: Facilitating MAT Acceptance & Implementation in Problem Solving & Felony Courts
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Development and Research Institutes, Inc. (Other)
Collaborators: Treatment Alternatives for Safe Communities (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NationalDRI; R34DA038799 (NIH)
Record Dates: First submitted 2017-07-14; First posted 2017-07-25 (Actual); Last update posted 2017-07-25 (Actual); Status verified 2017-07

CONDITIONS: Improving Treatment for Opioid Use Disorder in Courts

STUDY DESIGN:
Intervention Model Description: This study will develop and test the feasibility of an interactive eLearning modality and an eLearning + an organizational approach (change team intervention; a Technology Transfer model) to advance knowledge and facilitate inclusion of MAT in the criminal justice system for opioid-addicted clients. Courts recruited for the study will receive eLearning and half of these courts will be randomly assigned to the change team.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- E-learning intervention (Active Comparator): The E-learning intervention consists of two 20-minute e-learning modules that combine a didactic component with testimonials from respected professionals in the fields of addiction treatment and criminal justice. Module 1 describes the nature of opioid addiction and treatment modalities. Module 2 addresses specific criminal justice concerns of cost, acceptance, usefulness, and diversion, perceived obstacles to providing MAT access as described to us by Ohio criminal justice professionals in formative phase. All courts recruited for the study are exposed to E-Learning.
  Interventions: Behavioral: eLearning Modules
- Change Team Intervention (Experimental): Half of the courts exposed to e-learning will be randomly assigned to a change team intervention. The change team will reinforce the information in the modules and provide instrumental assistance in linking courts to MAT providers and financial resources.
  Interventions: Behavioral: eLearning Modules; Behavioral: Change Team Intervention

INTERVENTIONS:
Behavioral: eLearning Modules — All participating courts will view two eLearning modules. Module one discusses opioid addiction and treatment; module two discusses specific concerns of criminal justice with regard to MAT and ways in which those concerns may be addressed.
Behavioral: Change Team Intervention — Courts selected for the experimental condition will participate in a hands-on change team intervention to provide instrumental assistance and to reinforce the information contained in the eLearning modules.
  Arms: Change Team Intervention

SUMMARY:
This study compares two methodologies for improving access to medication assisted treatment (MAT) in Ohio courts where MAT is currently restricted or prohibited. All participating courts are asked to view two educational modules. Module 1 addresses the nature of opioid addiction and treatment. Module 2 addresses concerns specific to criminal justice such as misuse and diversion of medications. Courts selected for the experimental group also receive a hands-on change team initiative in which specially trained professionals work with court staff to provide education and instrumental assistance in order to improve access to MAT for court supervisees who are opioid-dependent.

DETAILED DESCRIPTION:
Although there is robust evidence for the efficacy of medication assisted treatment (MAT), e.g., buprenorphine, extended-release naltrexone, methadone, this evidence-based treatment (EBT) is not available for the majority of opioid dependent clients (ODCs) in the criminal justice (CJ) population.

In a recent survey of drug courts our group found that less than half include MAT as a treatment option for their ODCs. Moreover among the minority of courts that do permit MAT, it is typically restricted. Responses by drug court personnel revealed serious concerns about diversion, misuse, and uncertainty about the efficacy of MAT, especially among courts in which MAT was unavailable. Despite these barriers, 70% of the courts indicated that with proper evidence MAT could be considered or expanded as a treatment option. To increase court professionals' understanding of MAT and facilitate decisions on whether MAT would be an appropriate treatment, we proposed a Stage I study to develop and test the feasibility of using an eLearning and an eLearning + a behavioral change team intervention, an Addiction Technology Transfer Center - ATTC - Technology Transfer [TT] model, to advance knowledge and facilitate inclusion of MAT as a treatment option in the criminal justice system (CJS) for ODCs. To enhance the eLearning modality we included testimonials from opinion leaders/early adopters of MAT (e.g., a drug court judge, a representative from the National Association of Drug Court Professionals, and treatment providers) who addressed specific concerns such as methods to identify qualified MAT providers, appraise treatment plans, and prevent and minimize negative effects of diversion and misuse. The behavioral change intervention will be based on a model of process improvement developed by the ATTC Network5 to expand treatment options for the management of opioid dependence, in this case MAT. The planned program represents the first study to: 1) include testimonials by opinion leaders in conjunction with an eLearning approach to spur inclusion of an evidence-based intervention for the treatment of opioid dependence within a criminal justice (CJ) setting and; 2) adapt the ATTC TT model to the specific goal of facilitating inclusion of MAT as a treatment option. Specific aims of the study are:

Aim 1. Develop an eLearning (web-based) intervention that will provide information about risks and benefits of MAT to help drug and felony court staff determine whether MAT is suitable for their clients. The protocol will include group discussions with both MAT-friendly and MAT-averse court personnel and inclusion of a MAT Advisory Panel (MAP), a team of experts in the implementation of MAT in CJ settings. Through an iterative process (review/revisions by MAT experts and court staff) we will develop a consensual outline representing topics that would be addressed by our web-based intervention. The objective will be to provide a balanced, thorough presentation of both benefits and risks of MAT provision and will specifically seek to address concerns about MAT provision such as diversion and misuse. Informed by diffusion of innovations theory, the eLearning modules will be enhanced by including testimony of criminal justice professionals about their experiences with MAT in their courtrooms, what their concerns had been prior to MAT adoption by their court, and how ￼these concerns (and other obstacles that emerged) were addressed.

￼ Aim 2. Develop a TT intervention to facilitate Courts' readiness and resources to engage in case-by-case inquiries to determine whether and under what circumstances to permit MAT. Working with ATTC TT experts we will develop a change team (CT) intervention for court representatives and treatment providers (including Judge, coordinator, administrator, and case-managers). The objective of the proposed CT intervention will be to: 1) Broker relationships between MAT providers and courts; ensuring that MAT providers will accept court referred individuals; 2) Reinforce the educational objectives - including addressing in substantive ways issues of availability, access (including cost), misuse, and diversion - with court personnel in order to expand policy and practice to include MAT; 3) Work with local MAT and other treatment providers to help create an environment in which MAT is accepted as part of the constellation of available treatments; 4) help develop protocols such as assertive ongoing monitoring and support to assure that MAT benefits are sustained once a client has been referred to treatment.

Aim 3. Conduct a small-scale trial to evaluate the preliminary effectiveness of the eLearning intervention, and the eLearning + change team intervention (TT-intervention). Targeting courts that either do not place their ODCs in MAT or tightly restrict MAT access, 24 courts will be randomly assigned to 1 of 2 treatment conditions: 1. Treatment as usual, followed by the eLearning intervention, or 2. eLearning intervention followed by the CT intervention. Outcomes include 1) the rate of enrollment of clients in MAT; 2) rate of referral of clients to MAT; 3) MAT Knowledge, 4) Willingness to use MAT, and 5) Barriers to MAT. We expect this development/pilot project will lead to a protocol to implement an EBT in the CJS; a setting with high numbers of ODCs.

ELIGIBILITY:
Inclusion Criteria:

* Over 18 years of age
* Court Personnel

Exclusion Criteria:

* Under 18 years of age
* Not employed by court

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 96 (Estimated)
Dates: Start 2016-04-15 (Actual); Primary Completion 2018-04 (Estimated); Study Completion 2018-04 (Estimated)

PRIMARY OUTCOMES:
Enrollment in Medication Assisted Treatment | 9 months
  Pre-post intervention comparison of enrollment in MAT among opioid-dependent supervisees. Using an online survey, investigators compare court-reported data for MAT enrollment.

SECONDARY OUTCOMES:
MAT referrals | 9 months
  Pre-post intervention comparison of referral to MAT for opioid-dependent supervisees. Using an online survey, investigators compare court-reported data for MAT referrals.
MAT knowledge/attitudes | 9 months
  Via online survey, MAT knowledge and attitude scale will be used to test pre-post changes in both knowledge of and attitudes toward MAT.
Willingness to refer clients to MAT | 9 months
  Courts asked how receptive they are to refer clients to MAT. Using an online survey, investigators ask judges to elaborate upon their willingness to refer clients to MAT.
Barriers to MAT | 9 months
  Courts complete a checklist of structural barriers such as cost, policy opposition, availability. Using an online survey, investigators compare court-reported data for barriers to MAT referral.

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Rosenblum, Principal Investigator — Executive Director
Locations (1):
- National Development and Research Institutes, Inc., New York, New York, United States

IPD SHARING:
Plan to Share IPD: No